CLINICAL TRIAL: NCT07044856
Title: The Effect of Distraction With the Help of Virtual Reality on Pain, Anxiety and Vital Signs in Patients Undergoing Lumbar Puncture
Brief Title: Effect of Virtual Reality Distraction on Pain, Anxiety, Vital Signs in Patients Undergoing Lumbar Puncture
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Nazan Tasan, master of science, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IU-HEM-NT-01
Record Dates: First submitted 2025-05-19; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Puncture; Virtual Reality; Distraction
Keywords: lumbar puncture; virtual reality; pain; anxiety; vital sings
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The study has a randomized controlled experimental study design.
Who Masked: Participant
Masking Description: Patients who will be included in the study will know which group they have been assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality experimental group (Experimental): Before the procedure, the patient's vital signs will be checked, and pain and anxiety will be assessed. This group will be shown a video using virtual reality glasses during the lumbar puncture procedure. After the intervention, the patient's vital signs will be checked again, and pain and anxiety will be assessed.
  Interventions: Behavioral: distraction with virtual reality
- control group (No Intervention): Before the procedure, the patient's vital signs will be checked and pain and anxiety will be assessed. No intervention will be made during the lumbar puncture procedure in this group. After the procedure, the patient's vital signs will be checked again and pain and anxiety will be assessed.

INTERVENTIONS:
Behavioral: distraction with virtual reality — Before the procedure, the patient's vital signs will be checked and pain and anxiety will be assessed. This group will be shown a video using virtual reality glasses during the lumbar puncture procedure. After the intervention, the patient's vital signs will be checked again and pain and anxiety will be assessed.
  Arms: virtual reality experimental group

SUMMARY:
Lumbar puncture (LP) is one of the most frequently applied interventional procedures in the clinical field. It is still used as the gold standard diagnostic tool in some infectious and non-infectious diseases. Its use in treatment also increases the clinical importance of lumbar puncture . Due to its wide range of indications, LP is a procedure that requires a professional approach in nursing care . Patients may feel anxious at every stage of the procedure. Pain and fear may be experienced due to the anesthesia procedure and needle movements during the procedure . Having to maintain the fetal position during the procedure may cause anxiety. This situation may result in deterioration in vital signs later on . Considering all these problems, this study was planned considering that distraction with the help of virtual reality in the nursing care of patients undergoing LP will have a positive effect on pain, anxiety and vital signs. The fact that there is no experimental study in the literature investigating the effect of virtual reality on pain, anxiety and vital signs during LP constitutes the strong and original aspect of the study. The aim of the study was to evaluate the effects of virtual reality on pain, anxiety and vital signs in patients undergoing lumbar puncture.

DETAILED DESCRIPTION:
Lumbar puncture (LP) is a procedure performed by entering the subarachnoid space through the lumbar 3-4 or lumbar 4-5 vertebral spaces for diagnosis and treatment. LP is indicated for the diagnosis of many diseases such as benign intracranial hypertension, subarachnoid hemorrhage, seizure disorders, cognitive disorders, movement disorders, abnormal radiological imaging, cancer-related diseases, fever, encephalitis, bacterial meningitis or multiple sclerosis, and for therapeutic applications such as intracranial pressure management . However, patients may experience the procedure as uncomfortable and sometimes painful . Pain during anesthesia, the patient having to hold their position (fetal position) fixed, the needle making waves in the CSF, and pain when the needle touches the nerves going to the leg or hip are among the situations that cause discomfort to the patient during LP . Whether for diagnostic or therapeutic purposes, the LP procedure can cause pain, fear and anxiety in patients . There have been different definitions of virtual reality since its first appearance. Zhang defined virtual reality as a virtual environment consisting of different sensory stimuli by combining computer software and hardware. Virtual reality used in health services has been defined as an interactive, entertaining and three-dimensional visual feedback treatment and education tool. Virtual reality studies have had different purposes and goals for their use in the health field. When the developed applications and studies are examined, virtual reality has been used for different purposes such as training of healthcare personnel, surgical simulations, auxiliary tools for treatment methods, and physical therapy simulations. In the literature, we come across studies where virtual reality is used to cope with situations that may have negative effects on the patient such as pain, anxiety, and fear that may occur due to medical procedures. Virtual reality applications have been successfully applied and positive results have been obtained in distracting attention, which is one of the non-pharmacological methods in pain management . There are no sufficient studies in the literature regarding the problems that the patient may encounter during the lumbar puncture procedure. Researchers' interest in studies focusing more on post-procedural complications may lead to neglecting the negative experiences experienced by patients during the procedure. Pain during anesthesia, fear related to the procedure, and anxiety related to the procedure are among the negative experiences experienced by patients during lumbar puncture. In order to better manage this process, nurses can keep the pain and anxiety under control during the procedure by distracting the patients and prevent deterioration of their vital signs. In parallel with the rapid advancement of technology, nursing science is also renewing itself and showing interest in current approaches. With virtual reality technology, patients are isolated from their sensory environment and transported to a new environment prepared for them. With this distraction method, the patient's perception of the procedure currently being performed decreases and their tolerance for negative experiences related to the procedure increases. This study was planned considering that virtual reality application would be effective in solving problems that may develop during lumbar puncture because it is simple, reliable, and inexpensive.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* 18 years of age and older
* No psychiatric problems
* No vision or hearing problems
* Able to communicate in Turkish
* No open wounds, cellulitis, infection or bleeding in the area where the application will be made
* No diagnosis of epilepsy, head and neck cancer or vertigo
* No acute or chronic pain

Exclusion Criteria:

* Individuals who have pain before the procedure and use any analgesic medication,
* Those who have chronic pain or anxiety disorder,
* Those who use anxiolytic and/or sedative medication,
* Those who do not agree to participate in the study will not be included in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Skala | The scale will be applied 15 minutes after the procedure
  It measures the intensity of pain in the patient. VAS is a scale with two different names on a 10 cm long vertical or horizontal line (0=no pain, 10=most severe pain). The patient is asked to mark the point on this line that corresponds to the intensity of pain he feels. The distance between the marked point and the lowest end of the line (0=no pain) is measured in centimeters and the numerical value found indicates the intensity of pain in the patient. An increase in the score obtained from the scale in the evaluation indicates an increase in pain.
State Anxiety Scale | The scale will be applied 15 minutes after the procedure
  The scale consists of the State Anxiety Scale, which determines how an individual feels at a certain moment and condition, and the Trait Anxiety Scale, which determines how an individual feels regardless of the situation and condition they are in. The State Anxiety Scale, which is structured to measure what is felt at that moment, will be used in this study. The State Anxiety Scale consists of 20 questions on a four-point Likert type. The expressions in the State Anxiety Scale are evaluated as none at all 1 point, a little 2 points, a lot 3 points, and completely 4 points. The scale score varies between 20-80, and an increase in the score obtained from the scale indicates an increase in the level of anxiety. A total of 0-19 points from the individual indicates no anxiety, 20-39 points indicate mild anxiety, 40-59 points indicate moderate anxiety, and 60-79 points indicate severe anxiety. It is stated that individuals who score above 60 on the State Anxiety Scale need professional help
Vital Signs Form | The scale will be applied 15 minutes after the procedure
  The Vital Signs Form, prepared by the researcher by scanning the literature, is a form in which the patient's vital signs (blood pressure, pulse, respiration, oxygen saturation) will be taken and recorded before and after the procedure.

SECONDARY OUTCOMES:
Virtual Reality Glasses Application Satisfaction Form | The scale will be applied 15 minutes after the procedure
  This form, prepared by the researcher by scanning the literature, consists of 3 questions planned to be applied to the experimental group after the intervention. Question 1: The satisfaction of the intervention group will be measured on a 10 cm long horizontal line with the help of VAS. (0=not satisfied at all, 10=very satisfied). The higher the score, the higher the satisfaction. Question 2 asks whether the intervention group would prefer virtual reality if a lumbar puncture were to be performed again. The answer is yes or no. The third question is the intervention group's question 'Would you recommend virtual reality to other patients who will undergo lumbar puncture?' The answer is given as yes or no.

CONTACTS AND LOCATIONS:
Locations (1):
- İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No